CLINICAL TRIAL: NCT03319654
Title: Impact of DNA Fragmentation in Sperm on Pregnancy Outcome After Intra-uterine Insemination in a Spontaneous Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Alessa Sugihara, ASugihara, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UZA TBM -DNA IUI 2017
Record Dates: First submitted 2017-09-15; First posted 2017-10-24 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Infertility Unexplained; Infertility, Male; DNA Damage
Keywords: Unexplained Infertility; Idiopathic Infertility; DNA damage; DNA fragmentation; Insemination
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Single center, university setting, no commercial affiliation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spontaneous cycle IUI (Experimental): DNA fragmentation by TUNEL assay
  DNA fragmentation will be measured both at the time of the diagnostic work-up as at the time of insemination.
  Interventions: Diagnostic Test: DNA fragmentation by TUNEL assay

INTERVENTIONS:
Diagnostic Test: DNA fragmentation by TUNEL assay — Direct DNA fragmentation testing with terminal deoxyuridine nick end labeling (TUNEL) assay.

SUMMARY:
Infertility affects about 10% of all couples and is defined by a failure to achieve a clinical pregnancy within a year of regular unprotected sexual intercourse. Up to one third of these couples will not have an identifiable cause after routine investigation, id est idiopathic infertility. The current diagnosis of male infertility relies on the World Health Organization (WHO) 2010 criteria which focus on concentration, motility and morphology in comparison to cut-off values of a fertile population. Alas, the relevance of the conventional semen analysis for the choice of treatment and the predictive value for an infertile couple with idiopathic or mild male infertility embarking on medically assisted reproduction (MAR) remains questionable. In other words, there is a strong clinical need to distinguish fertile from infertile men through new sperm function testing and to be able to select both the patient population who will benefit from MAR as well as the type of treatment.

Numerous studies utilizing different techniques for assessing sperm DNA fragmentation support the existence of a significant association between sperm DNA damage and pregnancy outcomes.

In this prospective cohort study the investigators aim to study the role of sperm DNA fragmentation analysis in selecting the patient who will benefit from intra-uterine insemination (IUI) therapy since IUI is still considered the first step in MAR and is performed at a large scale in Belgium and worldwide.

ELIGIBILITY:
Inclusion Criteria:

Couples seeking fertility treatment after at least 12 months of unprotected intercourse are eligible. All couples underwent basic fertility investigations which included semen analysis, evaluation of menstrual cycle, and tubal patency testing.

Exclusion Criteria:

Double sided tubal disease, severe endometriosis (classified as revised American Society for Reproductive Medicine stage III or IV), premature ovarian failure, and known endocrine disorders (such as Cushing's syndrome or adrenal hyperplasia), azoö- or necrozoospermia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessa N Sugihara, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Sugihara A, Punjabi U, Roelant E, De Neubourg D. Is There a Relationship between Sperm DNA Fragmentation and Intra-Uterine Insemination Outcome in Couples with Unexplained or Mild Male Infertility? Results from the ID-Trial. Life (Basel). 2022 Dec 20;13(1):11. doi: 10.3390/life13010011. PMID 36675960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Centre for Reproductive Medicine of the Antwerp University Hospital, Belgium
Pre-assignment Details: 6 included patients did not proceed to treatment; 1 due to spontaneous pregnancy - 5 loss to follow-up
Groups:
- Spontaneous Cycle IUI: DNA fragmentation by TUNEL assay
  DNA fragmentation will be measured both at the time of the diagnostic work-up as at the time of insemination.
  DNA fragmentation by TUNEL assay: Direct DNA fragmentation testing with terminal deoxyuridine nick end labeling (TUNEL) assay.
Period: Overall Study
Arm/Group | Spontaneous Cycle IUI
Started | 114 (The couples underwent natural cycle IUI with or without ovulation trigger until pregnancy was achieved for a maximum of four cycles.)
Completed | 114
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since this study relates to fertility, we have included "couples". 114 couples were included hence 114 women and 114 men.
Groups:
- Spontaneous Cycle IUI: The couples underwent natural cycle IUI with or without ovulation trigger until pregnancy was achieved for a maximum of four cycles.
  DNA fragmentation was measured by TUNEL assay.
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 228
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 114 couples were included
  years
    Women: number analyzed (Participants) | 114
    Women | 30.3 (3.7)
    Men: number analyzed (Participants) | 114
    Men | 32.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 114
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Infertility Duration [Mean (Standard Deviation); unit: months] | 23.3 (12.4)
Sperm concentration [Median (Standard Deviation); unit: Million spermatozoa /ml ejaculate] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  Million spermatozoa /ml ejaculate
    number analyzed (Participants) | 113
    (all) | 48 (63.7)
Sperm progressive motility [Median (Standard Deviation); unit: % progessively motile spermatozoa] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  % progessively motile spermatozoa
    number analyzed (Participants) | 113
    (all) | 55 (16)
Abstinence period [Median (Standard Deviation); unit: days] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  days
    number analyzed (Participants) | 113
    (all) | 4 (2)
Semen volume [Median (Standard Deviation); unit: ml ejaculate] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  ml ejaculate
    number analyzed (Participants) | 113
    (all) | 3.7 (2.3)
Total sperm count [Median (Standard Deviation); unit: Million spermatozoa] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  Million spermatozoa
    number analyzed (Participants) | 113
    (all) | 165.2 (199)
Sperm ideal morphology [Median (Standard Deviation); unit: % of total sperm count] — Population: This pertains to 113 men (out of the 114 included). Rarely, patients did not have a diagnostic sperm analysis at our center but elsewhere.
  % of total sperm count
    number analyzed (Participants) | 113
    (all) | 5 (5)
% SDF total in ejaculate [Median (Standard Deviation); unit: % of spermatozoa with SDF in ejaculate] — Sperm DNA fragmentation measured by TUNEL in the total sperm population of the ejaculate Population: 104 men had a diagnostic sperm analysis with measurement of Sperm DNA fragmentation.
  % of spermatozoa with SDF in ejaculate
    number analyzed (Participants) | 104
    (all) | 9 (7.2)
% SDF vital in ejaculate [Median (Standard Deviation); unit: % of vital sperm with SDF in ejaculate] — Sperm DNA fragmentation measured by TUNEL in the vital sperm population of the ejaculate Population: 104 men had a diagnostic sperm analysis with measurement of Sperm DNA fragmentation.
  % of vital sperm with SDF in ejaculate
    number analyzed (Participants) | 104
    (all) | 1 (0.9)
Mean menstrual cycle length [Mean (Standard Deviation); unit: days] — Population: Data available of 111 out of 114 included wommen
  days
    number analyzed (Participants) | 111
    (all) | 29 (2)

OUTCOME MEASURES:

1. Primary Outcome: DNA Fragmentation as a Predictor of Live Birth Rate
Description: The odds ratio on live birth per unit increase in % total Sperm DNA Fragmentation of the diagnostic sample.
Time Frame: up to 36 months
Measure: Count of Participants; unit: Participants
Groups:
- Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis: 114 couples underwent natural cycle IUI with or without ovulation trigger until pregnancy was achieved for a maximum of four cycles.
Arm/Group | Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis
Number analyzed (Participants) | 114
Participants | 32
Statistical Analysis 1: Comparison: Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis; The null hypothesis is: there is no association between % total Sperm DNA Fragmentation and live birth; Test type: Other — A generalized estimating equation (GEE)-model with an exchangeable correlation structure and a logit link function was used to analyze the probability of live birth and clinical pregnancy respectively. All IUI cycles are used in this model with correction for the fact that cycles of the same couple are not independent; p = 0.04, GEE-model; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.90 to 0.9985]
Statistical Analysis 2: Comparison: Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis; Test type: Other; p > 0.05, Receiver Operating Characteristics curve; Area under the ROC curve = 0.576

2. Secondary Outcome: % SDF in the Total Fraction After Density Gradient in the Diagnostic Sample (Pre-IUI)
Description: % of spermatozoa with DNA fragmentation in the total fraction after density gradient in the diagnostic sample (pre-IUI)
Time Frame: up to 3 months
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Groups:
- Spontaneous Cycle IUI: DNA fragmentation by TUNEL assay after density gradient (diagnostic sample)
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 102
% of spermatozoa with SDF | 9.6 [4.6 to 20.1]

3. Secondary Outcome: % SDF in the Vital Fraction After Density Gradient in the Diagnostic Sample (Pre-IUI)
Description: % of spermatozoa with DNA fragmentation in the vital fraction after density gradient in the diagnostic sample (pre-IUI)
Time Frame: up to 3 months
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 102
% of spermatozoa with SDF | 0.6 [0.2 to 1]

4. Secondary Outcome: % SDF in the Total Fraction in the Ejaculate of the IUI- Sample
Description: % of spermatozoa with DNA fragmentation in the total fraction in the ejaculate (before density gradient) of the IUI-sample
Time Frame: 36 months
Population: number of semen samples for IUI analyzed for sperm DNA fragmentation before density gradient
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Groups:
- Spontaneous Cycle IUI: DNA fragmentation by TUNEL assay before density gradient (IUI sample)
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 209
% of spermatozoa with SDF | 8 [5 to 12]

5. Secondary Outcome: % SDF in the Vital Fraction in the Ejaculate of the IUI- Sample
Description: % of spermatozoa with DNA fragmentation in the vital fraction in the ejaculate (before density gradient) of the IUI-sample
Time Frame: 36 months
Population: number of semen samples for IUI analyzed for sperm DNA fragmentation before density gradient
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 209
% of spermatozoa with SDF | 1 [0 to 2]

6. Secondary Outcome: % SDF in the Total Fraction After Density Gradient in the IUI Sample
Description: % of spermatozoa with DNA fragmentation in the total fraction after density gradient in the IUI sample
Time Frame: 36 months
Population: number of semen samples for IUI analyzed for SDF after density gradient
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Groups:
- Spontaneous Cycle IUI: DNA fragmentation by TUNEL assay after density gradient (IUI sample)
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 210
% of spermatozoa with SDF | 8.3 [4 to 14]

7. Secondary Outcome: % SDF in the Vital Fraction After Density Gradient in the IUI Sample
Description: % of spermatozoa with DNA fragmentation in the vital fraction after density gradient in the IUI sample
Time Frame: 36 months
Population: number of semen samples for IUI analyzed for SDF after density gradient
Measure: Median (Inter-Quartile Range); unit: % of spermatozoa with SDF
Arm/Group | Spontaneous Cycle IUI
Number analyzed (Participants) | 210
% of spermatozoa with SDF | 0.4 [0.2 to 1]

ADVERSE EVENTS:
Time Frame: 36 months.
Description: This was a non-interventional study. SDF testing was only carried out when the inseminating motile count was deemed sufficient, as such the treatment would not be jeopardized.
  The result of the SDF test did not interfere with the allocated treatment.
Groups:
- Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis: 114 couples underwent natural cycle IUI with or without ovulation trigger until pregnancy was achieved for a maximum of four cycles.
  Sperm DNA fragmentation testing was carried out on the diagnostic and IUI samples.
Arm/Group | Spontaneous Cycle IUI - Sperm DNA Fragmentation Analysis
All-Cause Mortality (participants affected / at risk) | 0/228
Serious Adverse Events (participants affected / at risk) | 0/228
Other Adverse Events (participants affected / at risk) | 0/228

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT03319654/Prot_SAP_000.pdf